CLINICAL TRIAL: NCT02383368
Title: An Open-Label, Dose-Escalation/Expansion Phase 1 Study of ASP4132 Given Orally to Patients With Advanced Refractory Solid Tumors and Lymphoma
Brief Title: A Dose Escalation and Expansion Study of ASP4132 to Subjects With Advanced Refractory Tumors and Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4132-CL-0001
Record Dates: First submitted 2015-03-04; First posted 2015-03-09 (Estimated); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Lymphoma; Refractory Solid Tumors; Advanced Cancer
Keywords: Pharmacokinetics; ASP4132; Lymphoma; Refractory Solid Tumors
MeSH Terms: conditions — Lymphoma | interventions — ASP4132

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ASP4132 dose escalation (Experimental): Subjects will receive a single dose of the study drug on Day -4 (Single-Dose Period), followed by PK sampling prior to Multiple-Dose Period where they will receive the same dose as they received in the Single-Dose Period on one of four schedules:
  Continuous - daily dosing for 28 days, Intermittent: Schedule A: 3 days on / 4 days off; Schedule B: 1 days on / 6 days off; Schedule C: 3 days on / 11 days off.
  Interventions: Drug: ASP4132
- ASP4132 dose expansion (Experimental): Subjects in Part 2 will be treated with ASP4132 at the MTD and dosing schedule identified from Part 1.
  Interventions: Drug: ASP4132

INTERVENTIONS:
Drug: ASP4132 — oral

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of ASP4132 and to determine the maximum tolerated dose and recommended phase 2 dose of ASP4132. The study will also determine the pharmacokinetics (PK) of ASP4132 and evaluate the preliminary antitumor activity.

DETAILED DESCRIPTION:
The study consists of two parts and these will be conducted sequentially: Part 1 (dose escalation) and Part 2 (dose expansion). Subjects will participate in Part 1 or Part 2.

ELIGIBILITY:
Inclusion Criteria:

* Subject has a life expectancy of more than 3 months
* Subject agrees not to participate in another interventional study while on treatment.
* Subject has an Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2.
* Female subject must be either:

  1. Of non-child bearing potential:

     * post-menopausal (defined as at least 1 year without any menses) prior to Screening,
     * or, documented surgically sterile or status post hysterectomy
  2. Or, if of childbearing potential,

     * agree not to try to become pregnant during the study and for 90 days after the final study drug administration;
     * if heterosexually active must use two forms of birth control
* Male subject and their female spouse/partners who are of childbearing potential must be using highly effective contraception consisting of two forms of birth control (one of which must be a barrier method) starting at Screening and continue throughout the study period and for 90 days after the final study drug administration.
* Subject must have advanced and/or metastatic, histologically or cytologically documented cancer or lymphomas, for whom there is no available standard therapy shown to provide clinical benefit.

Exclusion Criteria:

* Subject has absolute neutrophil count < 1000/μL, platelet count < 75,000/μL, and hemoglobin < 8 g/dL (< 5 mmol/L) at Screening
* Subject has total serum bilirubin ≥1.5 times the upper limit of normal (ULN),serum alanine aminotransferase (ALT), aspartate aminotransferase (AST) > 3 times ULN, or albumin ≤ 3.0 g/dL at Screening.
* Subject has any abnormalities in serum sodium, potassium, chloride, calcium and magnesium levels ≥ Grade 2 at screening (CTCAE Version 4.03).
* Subject has a known elevation in serum lactate at screening ˃ 2x institutional ULN
* Subject has an estimated glomerular filtration rate (eGFr) of < 60ml/min as calculated by the modification of diet Renal disease (MDRD) Equation.
* Subject with a QTcF of > 450 msec in male subjects and > 470 msec in female subjects on the screening 12 lead ECG.
* Subject has Neuropathy ≥ Grade 2 at Screening.
* Subject has Type 1 Diabetes Mellitus or Type 2 Diabetes Mellitus and currently being treated with insulin or sulfonylureas.
* Subject has concomitant active second malignancies unless remission was achieved at least 3 years prior to study entry and subject is no longer on therapy for the malignancy.
* Subject has a significant cardiovascular disease
* Subject has a known history of acute or chronic hepatitis B (HBV), HIV or hepatitis C (HCV) infection.
* Subject has serious/active bacterial, viral or fungal infection requiring systemic treatment.
* Subject has significant gastrointestinal abnormalities, including ulcerative colitis, chronic diarrhea associated with intestinal malabsorption, Crohn's disease, and/or prior surgical procedures affecting absorption or requirement for intravenous (IV) alimentation.
* Subject has active central nervous system (CNS) metastases not controlled by prior surgery or radiotherapy (subjects must be off steroids). Subjects with signs or symptoms suggestive of brain metastasis are not eligible unless brain metastases are ruled out by brain MRI/CT.
* Subject has concurrent severe or uncontrolled medical disease or organ system dysfunction which, in the opinion of the Investigators, would limit life expectancy to < 3 months.
* Subject has psychiatric disorder or altered mental status that would preclude an understanding of the informed consent process and/or completion of the necessary study procedures.
* Subject has difficulty swallowing large pills.
* Subject currently being treated with biguanides or other agents known to increase risk of lactic acidosis.
* Subject has unavoidable concomitant treatment with any drug known for causing Torsades de Pointes.
* Subject has had radiotherapy or surgery within the 4 weeks prior to treatment with ASP4132.
* Subject has not discontinued all previous systemic therapies for cancer including chemotherapy, immunotherapy, or biological therapies for at least 14 days prior to the initiation of ASP4132.
* Subject has not fully recovered from the acute toxicities (except alopecia) of any prior anti-cancer therapy.
* Subject requiring concomitant use of strong CYP3A4 inhibitors or inducers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2015-03-23 (Actual); Primary Completion 2018-04-27 (Actual); Study Completion 2018-04-27 (Actual)

PRIMARY OUTCOMES:
Safety as assessed by adverse events | up to 39 months
Safety as assessed by clinical laboratory tests | up to 39 months
Safety as assessed by vital signs | up to 39 months
Safety as assessed by electrocardiograms (ECG) | up to 39 months

SECONDARY OUTCOMES:
Objective response rate to ASP4132 | Week 16
Duration of response to ASP4132 | Week 16
Disease control rate to ASP4132 | Week 16
Maximum concentration (Cmax) of ASP4132 | up to 43 days
Time of the maximum concentration (Tmax) of ASP4132 | up to 43 days
Area under the concentration-time curve from time of dosing to the last measurable concentration (AUClast) of ASP4132 | up to 43 days
AUC from the time of dosing to 24 hours (AUC24) of ASP4132 | up to 43 days
AUC from the time of dosing extrapolated to time infinity (AUCinf) of ASP4132 | up to 43 days
Apparent terminal elimination half-life (T1/2) of ASP4132 | up to 43 days
Accumulation ratio of ASP4132 | up to 43 days
Apparent total systemic clearance after single or multiple extravascular dosing (CL/F) of ASP4132 | up to 43 days
Apparent volume of distribution during the terminal elimination phase after single or multiple extravascular dosing (Vz/F) of ASP4132 | up to 43 days
Progression-free survival | up to 39 months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Global Development, Inc.
Locations (5):
- United States (5):
  - Site US10001, New Haven, Connecticut
  - Site US10004, Chicago, Illinois
  - Site US10002, Rochester, Minnesota
  - Site US10003, Houston, Texas
  - Site US10005, Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- [Derived] Janku F, LoRusso P, Mansfield AS, Nanda R, Spira A, Wang T, Melhem-Bertrandt A, Sugg J, Ball HA. First-in-human evaluation of the novel mitochondrial complex I inhibitor ASP4132 for treatment of cancer. Invest New Drugs. 2021 Oct;39(5):1348-1356. doi: 10.1007/s10637-021-01112-7. Epub 2021 Apr 8. PMID 33830407
- See also: Link to results on the Astellas Clinical Study Results website — https://astellasclinicalstudyresults.com/study.aspx?ID=316